CLINICAL TRIAL: NCT00248885
Title: Peri-Operative Morbidity and Quality of Life After CABG
Brief Title: Peri-Operative Morbidity and Quality of Life After Coronary Artery Bypass Graft (CABG)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Mary E. Charlson, Weill Cornell. Medical College
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 0001004169 (Formerly 0100-006)
Record Dates: First submitted 2005-11-03; First posted 2005-11-04 (Estimated); Last update posted 2008-04-11 (Estimated); Status verified 2008-04

CONDITIONS: Coronary Artery Bypass Graft Surgery
Keywords: Coronary artery bypass graft surgery; Perioperative complications; Neurocognitive function; Quality of life; Blood pressure

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): In this group (Low) the goal was to maintain MAP between 50-60 mm Hg during CPB.
  Interventions: Procedure: Regulating Mean Arterial Pressure during cardiopulmonary bypass
- 2 (Experimental): In this group (High), the goal was to maintain MAP between 80-100 mm Hg during CPB.
  Interventions: Procedure: Regulating Mean Arterial Pressure during cardiopulmonary bypass

INTERVENTIONS:
Procedure: Regulating Mean Arterial Pressure during cardiopulmonary bypass — Patients were randomized to one of two groups. In the first group (Low) the goal was to maintain MAP between 50-60 mm Hg during CPB. In the second group (High), the goal was to maintain MAP between 80-100 mm Hg. In both groups, CPB flow was held constant at 1.6 L/min/M2 (cool) and 2.4 L/min/M2 (warm) and vasoactive drugs (nitroglycerin or phenylephrine) were used to maintain MAP in the desired range. MAP was controlled in this fashion from the onset of CPB through separation from CPB began.
  Other Names: Mean Arterial Pressure during cardiopulmonary bypass 50-60 mm/Hg (control) vs. 80-100 mm/Hg (experimental)

SUMMARY:
It is the long term objective of this study to preserve or improve the quality of life and to prevent deterioration in physical and mental function following myocardial revascularization among bypass surgery patients.

DETAILED DESCRIPTION:
The objective of this study is to compare the efficacy of two strategies of intra-operative hemodynamic management in preventing peri-operative cardiac, cognitive and neurologic morbidity and mortality and postoperative deterioration in the patient's quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. Patients had to be undergoing elective CABG, without concomitant valve or other cardiac surgery.
2. Patients also had to be able to perform the neuropsychologic tests, and to provide informed consent.

Exclusion Criteria:

1. Patients who refused to participate in the study.
2. Patients who live too far away from NYC to be able to come back for follow up at six months post-operatively.
3. Patients who had either valvular replacement and aortic amd mitral an aneurysm repair, or other cardiothoracic surgery.
4. Patients who were unable to complete the neuropsychologic test.
5. Patient who were part of another CABG study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 248 (Actual)
Dates: Start 1991-09; Study Completion 1994-09 (Actual)

PRIMARY OUTCOMES:
Cardiac morbidity | 6-months after surgery
Neurologic morbidity | 6-months after surgery
Mortality | 6-months after surgery
Functional status | 6-months after surgery
Neurocognitive function | 6-months after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Mary E Charlson, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- New York Presbyterian Hospital-Weill Cornell Medical College, New York, New York, United States